CLINICAL TRIAL: NCT05602571
Title: Effects of Adding Platelet-Rich Plasma (PRP) Therapy to Extracorporeal Shock Wave Therapy (ESWT) in Patients With Lateral Epicondylitis: Double-Blind Randomized Sham-Controlled Study
Brief Title: The Effectiveness of the Combination of PRP and ESWT in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Ali İzzet Akçin, Principal Investigator-Research Assistant-MD, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEPRPESWT22
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Musculoskeletal Diseases; Elbow Tendinitis; Lateral Epicondylitis; Platelet-Rich Plasma (PRP)
Keywords: Lateral Epicondylitis; Extracorporeal Shockwave Therapy (ESWT); Platelet-Rich Plasma (PRP)
MeSH Terms: conditions — Musculoskeletal Diseases; Tennis Elbow

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT+Exercise (Experimental): Home exercise program including stretching and eccentric strengthening exercises twice a day for 3 months + 3 sessions of ESWT once a week for 3 weeks.
  Interventions: Other: ESWT+Exercise
- PRP+ESWT+Exercise (Active Comparator): Home exercise program including stretching and eccentric strengthening exercises twice a day for 3 months + 3 sessions of ESWT once a week for 3 weeks + PRP injection
  Interventions: Procedure: PRP+ESWT+Exercise
- Sham PRP+ESWT+Exercise (Sham Comparator): Home exercise program including stretching and eccentric strengthening exercises twice a day for 3 months + 3 sessions of ESWT once a week for 3 weeks + Sham PRP injection
  Interventions: Procedure: Sham PRP+ESWT+Exercise

INTERVENTIONS:
Other: ESWT+Exercise — Radial ESWT treatment will be applied to patients for 3 weeks, once a week for a total of 3 sessions. Radial shock waves will be applied in circular motions by applying gel on the epicondylar area where the most pain and sensitivity is. In each session, 8 Hz, 2.0 bar, 2000 beats will be applied.
  Therapeutic Exercise:
  All patients will be taught a home exercise program including stretching and eccentric strengthening exercises by an experienced physiotherapist. The eccentric exercises consisted of the following: three sets of 10 repetitions for wrist and elbow ﬂexion; two sets of 10 repetitions for wrist extension strengthening, starting with 50% of maximum strength and density and increasing the resistance each week; and ﬁnally, two sets of 10 repetitions for the wrist ﬂexor and extensor muscle groups comprising 20s of stretching and 10s of relaxing using the unaﬀected hand. Exercise program will be done twice a day for 3 months.
  Arms: ESWT+Exercise
Procedure: PRP+ESWT+Exercise — Radial ESWT treatment will be applied to patients for 3 weeks, once a week for a total of 3 sessions. Radial shock waves will be applied in circular motions by applying gel on the epicondylar area where the most pain and sensitivity is. In each session, 8 Hz, 2.0 bar, 2000 beats will be applied.
  Therapeutic Exercise:
  All patients will be taught aforementioned home exercise program. Exercise program will be done twice a day for 3 months.
  Procedure:
  10 ml of venous blood taken from the patients will be put into the T-LAB® PRP kit (T-Biotechnology Laboratory, İstanbul, Turkey) and will then be centrifuged. Approximately 3 cc of the PRP obtained will be applied to the tendinosis area under USG guidance. All injections will be performed with long axis in-plane technique, using the ultrasound device (Esaote My Lab 70 XVision 6-18 Mhz linear probe).
  Arms: PRP+ESWT+Exercise
Procedure: Sham PRP+ESWT+Exercise — Radial ESWT treatment will be applied to patients for 3 weeks, once a week for a total of 3 sessions. Radial shock waves will be applied in circular motions by applying gel on the epicondylar area where the most pain and sensitivity is. In each session, 8 Hz, 2.0 bar, 2000 beats will be applied.
  Therapeutic Exercise:
  All patients will be taught aforementioned home exercise program. Exercise program will be done twice a day for 3 months.
  Procedure:
  In Sham-PRP group,10 ml of venous blood will be taken and after the same waiting time 3 cc of 0.9% saline will be injected to the tendinosis area under USG guidance. All injections will be performed with long axis in-plane technique, using the ultrasound device (Esaote My Lab 70 XVision 6-18 Mhz linear probe).
  Arms: Sham PRP+ESWT+Exercise

SUMMARY:
The aim of this study is to determine the effectiveness of adding PRP or Sham PRP injection to ESWT treatment in patients with lateral epicondylitis on pain, muscle strength, functional activities, quality of life and work activities, and to determine the superiority of the treatments over each other.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE) is one of the most common elbow problems. It is characterized by pain in the lateral epicondyle of the humerus and on the surface of the extensor muscles of the forearm. It is seen in those who perform activities involving repetitive forced wrist extension and can lead to chronic pain syndrome.

Various treatment methods are used in the treatment of LE in order to reduce the patient's pain and increase his/her functional capacity. There are more than 40 treatment methods in the literature such as oral and local non-steroidal anti-inflammatory drugs (NSAID), cold application, deep friction massage, stretching and strengthening exercises, ultrasound, laser, ESWT, corticosteroid/botulinum toxin/glucosamine/autologous blood/platelet rich plasma (PRP) injections, prolotherapy, acupuncture, manipulation, and surgery.

Extracorporeal shock wave therapy (ESWT) is a method that aims to provide treatment by focusing high amplitude sound waves on the area of the body to be applied.

PRP is an autologous concentration of human platelets in a small volume of plasma produced by centrifuging a patient's own blood.

This study was designed as a double-blind, prospective, placebo-controlled, randomized study. Participants were randomized into 3 groups: ESWT + therapeutic exercise, ESWT + Sham PRP injection + therapeutic exercise, ESWT + PRP injection + therapeutic exercise.

Visual Pain Scale (VAS), Patient Rated Tennis Elbow Evaluation (PRTEE), Quick Disabilities of the Arm, Shoulder and Hand Score (Quick DASH), SF (Short form) -36 Quality of Life Scale, Handgrip strength with Jamar hydraulic hand dynamometer, Common extensor tendon thicknesses, peritendinous fluid, bone irregularities, calcifications, and diffuse tendon heterogeneity with ultrasound, upper extremity muscle strength with Isomed 2000 isokinetic device will be evaluated.

It was planned that the evaluations were made and recorded by a blinded physician to the groups at the beginning of the treatment, at the 4th week and at the 12th week controls.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with lateral epicondylitis after physical examination
2. No other pathology detected on direct radiography
3. Complaints persisting for more than 3 months despite the application of other conservative treatment methods
4. Patients accepting to give blood for PRP or sham injection and can tolerate elbow injection and extracorporeal shock wave therapy (ESWT)

Exclusion Criteria:

1. Not being able to fully cooperate with the study and inability to read and write,
2. Injection (corticosteroid, PRP, etc.) treatment applied to the elbow area within three months,
3. Previous surgery or ESWT treatment in the area to be treated,
4. Pregnant women,
5. Arthritis (rheumatoid arthritis, spondyloarthritis, crystal arthropathies),
6. Those who have a history of direct trauma to the elbow and a history of fracture,
7. Those with a history of malignancy,
8. Bleeding diathesis,
9. Complex regional pain syndrome,
10. Presence of acute systemic infection,
11. Presence of local infection at the injection site,
12. Peripheral vasculopathy,
13. Cervical radiculopathy,
14. Patients with contraindications to ESWT application (pregnancy, cancer, coagulation disorders, inflammatory disease, pacemaker, metal implant in the area to be applied) were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline visual analog scale (VAS) elbow pain at 4th and 12th week | baseline and 12th week
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity. The patient will be asked to score rest, movement, and nighttime pain.

SECONDARY OUTCOMES:
Change from baseline Handgrip strength at 4th and 12th week | baseline and 12th week
  Measuring hand grip strength is an objective method for evaluating response to treatment and functional recovery. Grip strength will be evaluated with the Jamar hydraulic hand dynamometer. Patients will be asked to squeeze with maximum force and each measurement will be made three times, and their averages will be recorded in kg. The dynamometer has a dual scale readout which displays isometric grip force from 0-90 kg. Higher scores means better grip strength.
Change from baseline Quick Disabilities of the Arm, Shoulder and Hand Score (Quick DASH) at 4th and 12th week | baseline and 12th week
  Quick DASH is a questionnaire that can be used to evaluate disability, activity restriction and work participation restriction caused by musculoskeletal problems involving the upper extremity. The QuickDASH tool uses a 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not able to do at all) from which the patient can mark an appropriate number corresponding to his/her severity/function level. According to the results of the Quick DASH questionnaire, a score between 0-100 is obtained from each section and a higher score indicates greater disability.
Change from baseline quality of life (Short Form 36 (SF-36)) at 4th and 12th weeks | baseline and 12th week
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health. Total score was between 0 (disability) and 100 (no disability). Every subgroup of the questionnaire has a score scale between 0 and 100. Every increase in the subgroup of SF-36 questionnaire, which is a positive scoring system, indicates increase in quality of life related to health.
Change from baseline Ultrasonographic examination at 4th and 12th weeks | baseline and 12th week
  Ultrasonographic examination will be made using the Esaote My Lab 70 XVision 6-18 Mhz linear probe. Before the treatment, patients will be evaluated for tendinosis of the common extensor tendon (extensor carpi radialis brevis, extensor carpi ulnaris, extensor digitorum, extensor digiti minimini tendons) by a physician experienced in the field of ultrasound, as gray scale and color Doppler activity.
Change from baseline upper extremity muscle strength with isokinetic device at 4th and 12th weeks | baseline and 12th week
  Isokinetic systems are complex systems used for both rehabilitation and patient evaluation. Isokinetic contraction; It is defined as contraction at a constant rate throughout the entire range of motion and at an equal rate at all angles of motion. Wrist extensor strength isokinetic strength assessment will be performed by a physiotherapist who is trained in using the isokinetic device (IsoMed 2000, isokinetic dynamometer, Germany) and has at least 5 years of experience.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran EYVAZ, MD, Principal Investigator — Afyonkarahisar Health Sciences University; Ali İzzet AKÇİN, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunduz R, Malas FU, Borman P, Kocaoglu S, Ozcakar L. Physical therapy, corticosteroid injection, and extracorporeal shock wave treatment in lateral epicondylitis. Clinical and ultrasonographical comparison. Clin Rheumatol. 2012 May;31(5):807-12. doi: 10.1007/s10067-012-1939-y. Epub 2012 Jan 27. PMID 22278162
- [Background] Alessio-Mazzola M, Repetto I, Biti B, Trentini R, Formica M, Felli L. Autologous US-guided PRP injection versus US-guided focal extracorporeal shock wave therapy for chronic lateral epicondylitis: A minimum of 2-year follow-up retrospective comparative study. J Orthop Surg (Hong Kong). 2018 Jan-Apr;26(1):2309499017749986. doi: 10.1177/2309499017749986. PMID 29320964
- [Background] Arirachakaran A, Sukthuayat A, Sisayanarane T, Laoratanavoraphong S, Kanchanatawan W, Kongtharvonskul J. Platelet-rich plasma versus autologous blood versus steroid injection in lateral epicondylitis: systematic review and network meta-analysis. J Orthop Traumatol. 2016 Jun;17(2):101-12. doi: 10.1007/s10195-015-0376-5. Epub 2015 Sep 11. PMID 26362783
- [Derived] Akcin AI, Eyvaz N, Dundar U, Toktas H, Yesil H, Eroglu S, Adar S. The Clinical Efficacy of Extracorporeal Shock Wave Therapy Combined With Platelet-Rich Plasma and Exercise for Lateral Epicondylitis: Prospective Randomized Sham-Controlled Ultrasonographic Study. Arch Phys Med Rehabil. 2025 Aug;106(8):1173-1182. doi: 10.1016/j.apmr.2025.01.420. Epub 2025 Jan 20. PMID 39842562